CLINICAL TRIAL: NCT03263520
Title: Impact of the Use of Nandrolone on the Treatment of Malnutrition Induced by Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Erasto Gaertner (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HEG03
Record Dates: First submitted 2017-08-15; First posted 2017-08-28 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Cachexia; Cancer
MeSH Terms: conditions — Cachexia; Neoplasms | interventions — Nandrolone Decanoate; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Randomization will be made at the time of study enrollment by , where patients randomly selected as even number will be included in group 1 and those selected as odd number in group 2Group 1 (G1): the patient will receive an application of anabolic nandrolone decanoate at a dose of 50 mg (males) and 25 mg (females), intra-muscular form, in the first and fifteenth days. In addition to the anabolic steroid, the patient will use corticosteroids (dexamethasone) at home at a dose of 4 mg daily for both sexes.
  Group 2 (G2): The patient will use corticosteroids (dexamethasone) at a dose of 4 mg daily.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The outcomes assessor and investigator does not have contact with the patient or care provider at the moment of randomization and the study purpose. The investigator just apply the bioelectrical impedance analysis and helps the patient about doubts on the Quality of Life questionnaire of EORTC ( QLQ-C30)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: nandrolone and corticosteroid (Experimental): the patient will receive an application of anabolic nandrolone decanoate at a dose of 50 mg (males) and 25 mg (females), intra-muscular form, in the first and fifteenth days. In addition to the anabolic steroid, the patient will use corticosteroids (dexamethasone) at home at a dose of 4 mg daily by mouth on the morning for both sexes for 30 days.
  Interventions: Drug: Nandrolone Decanoate
- Group 2: corticosteroid (Active Comparator): Patient will take corticosteroids ( 4 mg of dexamethasone) per oral, QD at morning for 30 days
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Nandrolone Decanoate — Drug administration
  Other Names: Dexamethasone
  Arms: Group 1: nandrolone and corticosteroid
Drug: Dexamethasone — Drug administration
  Arms: Group 2: corticosteroid

SUMMARY:
Compare the use of nandrolone associated with corticosteroid for the treatment of cancer-induced malnutrition to treatment with corticosteroids alone in patients with tumors in the high gastro-intestinal tract, liver, pancreas and bile ducts in palliative treatment.

DETAILED DESCRIPTION:
* Compare muscle mass values obtained before and after the use of anabolic steroids upon assessment by bioelectrical impedance analysis (BIA).
* Compare the anabolic effect on quality of life (QLo) of the patient before and after the use of anabolic steroids.
* Compare data from laboratory tests such as complete blood count, albumin, C reactive protein and transferrin with drug intervention.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients above 18 years old.
* Patients with tumors in the high gastro-intestinal, hepatobiliary and pancreatic tracts in palliation.
* Patients able to undergo BIA.
* Malnourished patients as per the subjective global assessment produced by the patient (ASG-PPP) and whose score is greater than nine.
* Patients who agree to participate in the study.

Exclusion Criteria:

* Patients with malignant tumors of other metachronous or synchronous location except nonmelanoma skin tumor
* Patients with chronic renal failure.
* Patients on diuretics, recent or chronic.
* Patients on appetite stimulants and anabolic agents.
* Patients using pacemakers, which can interfere with the results of BIA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Compare the use of nandrolone associated with corticosteroid for the treatment of cancer-induced malnutrition to treatment with corticosteroids alone in cancer patients | After 30 days, the values will be compared to those obtained on the first consultant.
  Evaluate the BMI ( body mass index)- the weight in kilograms and the height in centimeters and BMI in Kg/ m2.
Compare the use of nandrolone associated with corticosteroid for the treatment of cancer-induced malnutrition to treatment with corticosteroids alone in cancer patients by bioimpedance analysis ( BIA) | After 30 days, the values will be compared to those obtained on the first consultant.
  Evaluate the BIA (biometrical impedance analysis)trough the reactance and resistance in ohms and the phase angle in degree.
ompare the use of nandrolone associated with corticosteroid for the treatment of cancer-induced malnutrition to treatment with corticosteroids alone in cancer patients trough quality of life assessment | After 30 days, the values will be compared to those obtained on the first consultant.
  Evaluate quality of life by European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnare Core 30 ( QLQ-C30), version 3.0 . The values are expressed as a percentage

SECONDARY OUTCOMES:
Compare data from laboratory tests: complete blood count, albumin, C reactive protein and transferrin with drug intervention. | After 30 days, the laboratory test will be collect again and the values will be compared to those obtained on the first consultant.
  The complete blood count will be expressed in millions by cubic milimiter( millions/mm3) , albumin in grams per deciliter (g/dL), C reactive protein in milligrams per deciliter (mg/dL), transferrin in milligrams per deciliter (mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Vinicius B Preti, MD, Principal Investigator — Hospital Erasto Gaertner/ Liga Paranaense de Combate ao Cancer
Locations (1):
- Hospital Erasto Gaertner, Curitiba, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: Undecided